CLINICAL TRIAL: NCT05838742
Title: A Multicentre Randomized, Double-blind, Placebo Controlled, Dose-finding, Phase 2 Study (MARS-17) of GSK3858279 in Adult Participants With Moderate to Severe Pain Due to Knee Osteoarthritis
Brief Title: A Dose-Finding Study to Evaluate the Efficacy and Safety of GSK3858279 in Adults With Knee Osteoarthritis (OA) Pain
Acronym: MARS-17
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study met futility criteria at pre-planned interim analysis, showing no clinical efficacy of the investigational drug. Based on the lack of efficacy at the interim data review, the sponsor decided to terminate the study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 209978; 2022-502799-22-00 (Other: EU-CT)
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Pain; Osteoarthritis, Knee
Keywords: Osteoarthritis; Musculoskeletal Diseases; 209978; GSK3858279; Efficacy; Safety; Pharmacokinetics
MeSH Terms: conditions — Pain; Osteoarthritis, Knee; Osteoarthritis; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- GSK3858279 - 60 mg weekly (Experimental): Participants received GSK3858279 60 milligram (mg) SC injection once per week for 16 weeks.
  Interventions: Drug: GSK3858279
- GSK3858279 - 240 mg every 2 weeks (Experimental): Participants received GSK3858279 240 mg SC injection every other week for 16 weeks. Placebo was given in the intervening week to maintain the blinding.
  Interventions: Drug: GSK3858279
- GSK3858279 - 240 mg weekly (Experimental): Participants received GSK3858279 240 mg SC injection once per week for 16 weeks.
  Interventions: Drug: GSK3858279
- GSK3858279 - 360 mg weekly (Experimental): Participants received GSK3858279 360 mg SC injection once per week for 16 weeks.
  Interventions: Drug: GSK3858279
- Placebo (Placebo Comparator): Participants received placebo subcutaneous (SC) injection once per week for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3858279 — GSK3858279 will be administered.
  Arms: GSK3858279 - 240 mg every 2 weeks; GSK3858279 - 240 mg weekly; GSK3858279 - 360 mg weekly; GSK3858279 - 60 mg weekly
Drug: Placebo — Placebo will be administered.
  Arms: Placebo

SUMMARY:
This is dose-finding study of GSK3858279 in participants with moderate to severe knee osteoarthritis pain. The purpose of this study is to investigate and provide the data necessary to select the optimal effective and safe dose(s) of GSK3858279.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 40 to 80 years of age inclusive
* OA of the index knee as defined by symptomatic for ≥ 6 months with a clinical diagnosis of OA as per American College of Rheumatology (ACR) clinical diagnosis criteria.
* Kellgren and Lawrence (KL) score ≥ 2 on X-ray in the index knee
* An average of the average daily pain score of ≥4 and less than or equal to (≤) 9 by the 11-point NRS (0-10)
* Body mass index (BMI) of < 40 kilogram per meter square (kg/m^2) (inclusive).
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular, renal, gastrointestinal, lymphatic disorders which in the opinion of the investigator would interfere with the study procedures and/or assessments.
* History or current evidence of any inflammatory arthritis such as rheumatoid arthritis, infective arthritis, Paget's disease, osteonecrosis, osteoporotic fracture, or any other joint disease that in the Investigator's opinion would interfere with the assessment of pain and other symptoms of osteoarthritis.
* History of significant trauma or surgery to a knee or hip within the last 6 months.
* Current immunodeficiency diseases including but not limited to acquired immunodeficiency disorder or immunoglobulin deficiency.
* Current or previous active Mycobacterium tuberculosis
* History or evidence of clinically significant multiple or severe drug allergies
* History of malignancy within the last 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Alanine transaminase (ALT) >1.5 times upper limit of normal (ULN).
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35 percent (%)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Evidence of renal insufficiency, indicated by estimated creatinine clearance < 60 milliliter/ minute (mL/min)/1.73 square meter (m^2) at screening.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (79):
- United States (14):
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Cooper City, Florida
  - GSK Investigational Site, Cutler Bay, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Williamsville, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Charlottesville, Virginia
- Argentina (6):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Buenos Aires-San Isidro
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires
  - GSK Investigational Site, Ciudad AutOnoma de Buenos Aire
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Mar del Plata
- Australia (4):
  - GSK Investigational Site, Botany, New South Wales
  - GSK Investigational Site, Kotara, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Camberwell, Victoria
- Canada (9):
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Guelph, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Winchester, Ontario
  - GSK Investigational Site, Joliette, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- China (11):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hohhot
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Shenyang
  - GSK Investigational Site, Shijiazhuang
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Zhuzhou
- France (5):
  - GSK Investigational Site, Dax
  - GSK Investigational Site, La Roche-sur-Yon
  - GSK Investigational Site, La Rochelle
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
- Germany (3):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Magdeburg
- Japan (7):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shimane
  - GSK Investigational Site, Tokyo
- Mexico (5):
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mexicali
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Torreón
- South Africa (4):
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Gauteng
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Stellenbosch
- GSK Investigational Site, Seoul, South Korea
- Spain (6):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
- United Kingdom (4):
  - GSK Investigational Site, Blackpool
  - GSK Investigational Site, Cannock
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 314 participants were enrolled in the study. Out of which 310 participants were included in the full analysis set (FAS) population.
Pre-assignment Details: Of 314 participants enrolled, 4 participants were randomized but did not receive study dose, hence were excluded from the FAS.
Period: Overall Study
Arm/Group | Placebo | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
Started (Randomized) | 107 | 51 | 51 | 52 | 53
Full Analysis Population | 105 | 50 | 51 | 51 | 53
Completed | 26 | 12 | 13 | 15 | 15
Not Completed | 81 | 39 | 38 | 37 | 38
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 3 | 3 | 1 | 4
Not completed — STUDY TERMINATED BY SPONSOR | 68 | 34 | 33 | 34 | 32
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0
Not completed — Randomized, not treated | 2 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set population included all randomized participants who received at least one dose of study intervention. Data was reported according to the randomized study intervention.
Groups:
- Placebo: Participants received placebo SC injection once per week for 16 weeks.
- GSK3858279 - 60 mg Weekly: Participants received GSK3858279 60 mg SC injection once per week for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly | Total
Number analyzed (Participants) | 105 | 50 | 51 | 51 | 53 | 310
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 63.7 (7.93) | 65.6 (9.11) | 63.6 (8.84) | 64.0 (8.99) | 64.5 (8.14) | 64.2 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 35 | 39 | 33 | 40 | 211
  Male | 41 | 15 | 12 | 18 | 13 | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 81 | 37 | 39 | 39 | 33 | 229
  Asian | 18 | 7 | 7 | 7 | 11 | 50
  Black or African American | 5 | 5 | 3 | 3 | 8 | 24
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 1 | 3
  Not reported | 1 | 1 | 1 | 0 | 0 | 3
  Unknown | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Average of Average Daily Knee Pain Intensity Using Numeric Rating Scale at Week 12
Description: Change from Baseline in knee pain due to Osteoarthritis were reported by weekly average of average daily pain numeric rating scale (NRS) at Week 12. The pain NRS is an 11-point scale (ranging from 0-10) for self-reporting of average daily knee pain where 0 indicates no pain, and 10 indicates the worst possible pain. For each participant, the weekly average of average daily pain score was calculated using the mean value of available daily pain scores falling in the assessment window for each week. A negative change from baseline indicates an improvement in pain. Participants were asked to complete the pain NRS questionnaire at the same time in the evening each day. Baseline scores were assigned based on an average of 7 days prior to day 1 dosing visit. Posterior mean change from baseline, 95 percent (%) credible interval (CI) was derived using Bayesian mixed model repeated measures. The data presented are the posterior mean with 95% confidence interval refers to 95% credible interval.
Time Frame: Baseline (Day -7 to Day -1) and at Week 12
Population: The analysis was performed on the full analysis set (FAS) that included all randomized participants who received at least one dose of study intervention. Only those participants who had a measured outcome used in estimation or imputed outcome based on composite intercurrent event strategy at the current time point were included in the overall number of participants analyzed field.
Measure: Mean (95% Confidence Interval); unit: Scores on Scale
Arm/Group | Placebo | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
Number analyzed (Participants) | 60 | 30 | 29 | 31 | 31
Scores on Scale | -2.13 [-2.55 to -1.73] | -1.66 [-2.24 to -1.10] | -1.88 [-2.46 to -1.31] | -1.74 [-2.32 to -1.17] | -2.03 [-2.60 to -1.47]
Statistical Analysis 1: Comparison: Placebo vs GSK3858279 - 60 mg Weekly; Test type: Other — Analysis performed using a Bayesian mixed model repeated measures adjusting for treatment, week, baseline, region and the treatment by week and baseline by week interactions using vague priors; Mixed Models Analysis; Analyzed using a joint model for change from baseline in average weekly pain score and time to intercurrent event handled using a composite strategy; Difference in Posterior Mean Change = 0.47, 95% CI 2-sided [-0.23 to 1.17]; Posterior mean difference with 95% credible interval is reported
Statistical Analysis 2: Comparison: Placebo vs GSK3858279 - 240 mg Every 2 Weeks; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in Posterior Mean Change = 0.25, 95% CI 2-sided [-0.46 to 0.95]; Posterior mean difference with 95% credible interval is reported
Statistical Analysis 3: Comparison: Placebo vs GSK3858279 - 240 mg Weekly; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in Posterior Mean Change = 0.39, 95% CI 2-sided [-0.31 to 1.10]; Posterior mean difference with 95% credible interval is reported
Statistical Analysis 4: Comparison: Placebo vs GSK3858279 - 360 mg Weekly; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in Posterior Mean Change = 0.11, 95% CI 2-sided [-0.60 to 0.80]; Posterior mean difference with 95% credible interval is reported

2. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score At Week 12
Description: The WOMAC pain subscale have a recall period of 48 hours and includes 5 subscales of pain assessment: 1-walking on flat, 2-going up downstairs, 3-at night while in bed, 4-sitting or lying; 5-standing upright. The total WOMAC pain subscale score ranges from 0-10; where 0 is no pain and 10 is extreme pain. The WOMAC pain subscale score was calculated by taking average of the 5 pain subscales at each visit. Change from baseline was calculated for each visit as the mean WOMAC Pain subscale score minus the mean baseline WOMAC Pain subscale score. A negative change from baseline indicates an improvement in pain. Baseline WOMAC scores for each participant were assigned based on the score measured prior to first dosing on Day1 visit. Posterior mean change from baseline, 95 percent (%) credible interval (CI) was derived using Bayesian mixed model repeated measures. The data presented are the posterior mean change from baseline with a 95% confidence interval refers to 95% Credible Interval.
Time Frame: Baseline (Day 1) and at Week 12
Population: The analysis was performed on FAS population which included all randomized participants who received at least one dose of study intervention. Only those participants who had a measured outcome used in estimation or imputed outcome based on composite intercurrent event strategy at the current time point were included in the overall number of participants analyzed field.
Measure: Mean (95% Confidence Interval); unit: Scores on Scale
Arm/Group | Placebo | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
Number analyzed (Participants) | 59 | 29 | 27 | 32 | 32
Scores on Scale | -2.16 [-2.59 to -1.74] | -2.13 [-2.73 to -1.52] | -2.21 [-2.82 to -1.59] | -1.95 [-2.54 to -1.36] | -1.93 [-2.52 to -1.36]

3. Secondary Outcome: Change From Baseline in WOMAC Physical Function Subscale Score at Week 12
Description: The WOMAC function subscale have a recall period of 48 hours and include 17 items of daily function assessments. The total WOMAC physical function subscale score ranges from 0-10 scale; where 0 is no difficulty and 10 is extremely difficult. The WOMAC physical function subscale score was calculated by taking the average of the 17 physical function subscales at each visit. Change from baseline was calculated for each visit as the mean WOMAC function subscale score minus the mean baseline WOMAC function subscale score. Baseline scores for each participant were assigned based on the score measured prior to first dosing on Day1 visit. A negative change from baseline indicated improvement. Posterior mean change from baseline, 95 percent (%) credible interval (CI) was derived using Bayesian mixed model repeated measures. The data presented are the posterior mean change from baseline with a 95% confidence interval refers to 95% Credible Interval.
Time Frame: Baseline (Day 1) and at Week 12
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Scores on Scale
Arm/Group | Placebo | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
Number analyzed (Participants) | 59 | 29 | 27 | 32 | 32
Scores on Scale | -1.94 [-2.36 to -1.53] | -1.99 [-2.58 to -1.40] | -1.56 [-2.15 to -0.97] | -1.65 [-2.23 to -1.08] | -1.65 [-2.22 to -1.11]

4. Secondary Outcome: Change From Baseline in Patient Global Assessment Of Disease (PtGA) at Week 12
Description: The PtGA is an assessment for disease conditions and intensity of knee osteoarthritis (OA) pain. Participants will respond on a Likert scale ranging from 1-5 based on the question "Considering all the ways in which your knee OA affects you, how do you feel your knee OA is doing today?" and to identify a number from 1 = very good (asymptomatic and no limitation to normal activities) to 5 = "very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher scores indicate worse conditions. Baseline scores for each participant were assigned based on the scores reported prior to first dosing on Day 1 visit. Posterior mean change from baseline, 95 percent (%) credible interval (CI) was derived using Bayesian mixed model repeated measures. The data presented are the posterior mean with a 95% confidence interval refers to 95% Credible Interval.
Time Frame: Baseline (Day 1) and at Week 12
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Scores on Scale
Arm/Group | Placebo | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
Number analyzed (Participants) | 58 | 28 | 27 | 32 | 32
Scores on Scale | -0.55 [-0.74 to -0.38] | -0.57 [-0.83 to -0.31] | -0.55 [-0.82 to -0.29] | -0.55 [-0.79 to -0.31] | -0.55 [-0.79 to -0.31]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs of Special Interest (AESI)
Description: AEs, SAEs, and AESIs were collected. An AE is any untoward medical occurrence in participant, temporally associated with use of study intervention, whether or not considered related to medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, medically important were categorized as SAEs. The AESIs of the study drug included serious and opportunistic infections, tuberculosis (TB) and TB reactivation, serious hypersensitivity reactions and Injection site reactions.
Time Frame: Up to 31 weeks
Population: The analysis was performed on safety population which included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
Number analyzed (Participants) | 105 | 50 | 51 | 51 | 53
Participants
  AEs | 69 | 29 | 32 | 32 | 34
  SAEs | 4 | 3 | 0 | 1 | 2
  AESIs | 14 | 3 | 4 | 2 | 12

6. Secondary Outcome: Number of Participants With Greater Than or Equal to (>=) Grade 3 Hematological/Clinical Chemistry Abnormalities According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCICTCAE)
Description: The laboratory measurements included hematology and clinical chemistry. The parameters evaluated were Basophil, Eosinophil, Erythrocyte Mean Corpuscular Hemoglobin, Erythrocyte Mean Corpuscular Volume, Erythrocytes, Hematocrit, Hemoglobin, Lymphocyte, Monocyte, Neutrophils, Platelets and Reticulocytes, Alanine Aminotransferase, Albumin, Alkaline phosphatase, Aspartate Aminotransferase, Bilirubin, Calcium, Creatinine, Direct Bilirubin, Glucose, Potassium, Sodium and Urea. Worst case grade (G) increase from baseline grade was provided for all the laboratory tests that were gradable by National Cancer Institute Common Terminology Criteria (NCI CTCAE, Version 5.0). Data for any participants with the worst-case grade changes (Increase or equal to Grade 3 or Increase to Grade 4) post-baseline are reported. Missing baseline grade was assumed as grade 0.
Time Frame: Up to 31 weeks
Population: The analysis was performed on safety population which included all participants who received at least 1 dose of study treatment. The overall number of participants analyzed represents only those participants available at the specified time points and evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
Number analyzed (Participants) | 99 | 48 | 48 | 47 | 49
Participants
  AST, Increase to Grade 3 | 0 | 0 | 0 | 1 | 0
  Creatine Kinase, Worsening to Grade 3 | 2 | 0 | 0 | 1 | 0
  Creatine Kinase, Worsening to Grade 4 | 0 | 0 | 1 | 1 | 0
  Gamma Glutamyl Transferase, Worsening to Grade 3 | 0 | 1 | 0 | 1 | 1
  Gamma Glutamyl Transferase, Worsening to Grade 4 | 1 | 0 | 0 | 0 | 0
  Lymphocyte count decreased, worsening to Grade 3: number analyzed (Participants) | 99 | 48 | 48 | 46 | 49
  Lymphocyte count decreased, worsening to Grade 3 | 0 | 1 | 0 | 0 | 0

7. Secondary Outcome: Maximum Concentration (Cmax) of GSK3858279
Description: Blood samples were collected at the indicated time points for pharmacokinetic (PK) analysis of GSK3858279 . Pharmacokinetic analysis was conducted using a model based analysis using all available data.
Time Frame: Pre-dose: Day 1, Weeks 1, 2, 4, 8, 10, 11 and 12
Population: The analysis was performed on PK set which included all randomized participants in the Safety Population who had at least 1 dose of GSK3858279 and at least 1 non-missing PK assessment (Non-quantifiable values were considered as non-missing values). Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
Number analyzed (Participants) | 26 | 23 | 25 | 25
nanograms/milliliter (ng/mL) | 4603.1 (48) | 12330.0 (47) | 15383.5 (51) | 22169.0 (40)

8. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of GSK3858279
Description: Tmax predicted from the population PK model fitted to GSK3859279 serum concentration time data collected at the indicated time points for PK analysis.
Time Frame: Pre-dose: Day 1, Weeks 1, 2, 4, 8, 10, 11 and 12
Population: as for outcome 7
Measure: Median (Full Range); unit: Day
Arm/Group | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
Number analyzed (Participants) | 26 | 23 | 25 | 25
Day | 1.454 [0.78 to 2.04] | 1.751 [0.94 to 3.90] | 1.412 [0.88 to 2.26] | 1.377 [0.73 to 2.26]

9. Secondary Outcome: Pre-Dose (Trough) Concentration at the End of the Dosing Interval (Ctau) of GSK3858279
Description: Ctau predicted from the population PK model fitted to GSK3859279 serum concentration time data collected at the indicated time points for PK analysis.
Time Frame: Pre-dose: Day 1, Weeks 1, 2, 4, 8, 10, 11 and 12
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
Number analyzed (Participants) | 26 | 23 | 25 | 25
ng/mL | 2449.9 (63) | 3076.6 (59) | 7224.0 (60) | 11037.5 (52)

10. Secondary Outcome: Average Concentration Over a Dosing Interval (Cavg) of GSK3858279
Description: Cavg predicted from the population PK model fitted to GSK3859279 serum concentration time data collected at the indicated time points for PK analysis.
Time Frame: Pre-dose: Day 1, Weeks 1, 2, 4, 8, 10, 11 and 12
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
Number analyzed (Participants) | 26 | 23 | 25 | 25
ng/mL | 3623.3 (51) | 7176.4 (48) | 11760.8 (53) | 16997.6 (42)

11. Secondary Outcome: Area Under the Time-Concentration Curve (AUC) Over the Dosing Interval (0-Tau) (AUC[0-Tau]) of GSK3858279
Description: AUC(0-tau) predicted from the population PK model fitted to GSK3859279 serum concentration time data collected at the indicated time points for PK analysis.
Time Frame: Pre-dose: Day 1, Weeks 1, 2, 4, 8, 10, 11 and 12
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
Number analyzed (Participants) | 26 | 23 | 25 | 25
day*ng/mL | 25362.8 (51) | 100469.4 (48) | 82325.8 (53) | 118983.5 (42)

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious adverse events (SAEs) and non-serious adverse events (Non-SAEs) were collected from the start of the study intervention (Day 1) until follow up of week 31.
Description: All-cause mortality, SAEs and Non-SAEs were reported for the Safety Population which included all randomized participants who received at least 1 dose of study treatment.
Arm/Group | Placebo | GSK3858279 - 60 mg Weekly | GSK3858279 - 240 mg Every 2 Weeks | GSK3858279 - 240 mg Weekly | GSK3858279 - 360 mg Weekly
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/50 | 0/51 | 0/51 | 0/53
Serious Adverse Events (participants affected / at risk) | 4/105 | 3/50 | 0/51 | 1/51 | 2/53
Other Adverse Events (participants affected / at risk) | 37/105 | 14/50 | 25/51 | 20/51 | 22/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=105) | GSK3858279 - 60 mg Weekly (N=50) | GSK3858279 - 240 mg Every 2 Weeks (N=51) | GSK3858279 - 240 mg Weekly (N=51) | GSK3858279 - 360 mg Weekly (N=53)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoedema (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=105) | GSK3858279 - 60 mg Weekly (N=50) | GSK3858279 - 240 mg Every 2 Weeks (N=51) | GSK3858279 - 240 mg Weekly (N=51) | GSK3858279 - 360 mg Weekly (N=53)
Nasopharyngitis (Infections and infestations) | 8 (8) | 2 (2) | 4 (4) | 4 (4) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (4) | 3 (5) | 2 (2) | 3 (4)
Headache (Nervous system disorders) | 10 (28) | 8 (14) | 10 (20) | 6 (8) | 5 (13)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (4) | 3 (4) | 1 (1) | 6 (7)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (6) | 2 (2) | 1 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (11) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Injection site reaction (General disorders) | 2 (5) | 1 (2) | 3 (14) | 1 (7) | 3 (5)
Injection site bruising (General disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Fatigue (General disorders) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (4) | 3 (4) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 4 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data do not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT05838742/Prot_004.pdf
  • Statistical Analysis Plan (2024-12-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT05838742/SAP_005.pdf